CLINICAL TRIAL: NCT05044949
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group Study Evaluating the Safety and Tolerability of Limosilactobacillus Reuteri Administered to Healthy Volunteers.
Brief Title: Study Evaluating the Safety and Tolerability of a Probioitc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CSUB0196
Record Dates: First submitted 2021-09-02; First posted 2021-09-16 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers; Tolerability; Safety
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose L reuteri capsules (Active Comparator): Subjects will be asked to consume 2 capsules with high dose L reuteri per day in 28 days.
  Interventions: Other: Probiotic
- High dose L reuteri capsules (Active Comparator): Subjects will be asked to consume 2 capsules with a low dose L reuteri per day in 28 days.
  Interventions: Other: Probiotic
- Placebo capsules (Placebo Comparator): Subjects will be asked to consume 2 capsules with placebo powder per day in 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic — The study product is a probiotic strain
  Arms: High dose L reuteri capsules; Low dose L reuteri capsules
Other: Placebo — The study product is a placebo to the probiotic strain
  Arms: Placebo capsules

SUMMARY:
The rationale for the current study is to initially evaluate the safety and tolerability of a novel strain of the probiotic Limosilactobacillus reuteri (L. reuteri) in healthy volunteers.

DETAILED DESCRIPTION:
Probiotics are live microorganisms, which when administered in adequate amounts, confer a health benefit on the host. Probiotics have been studied for decades for their potential health benefits of non-pathogenic microorganisms. The species Limosilactobacillus reuteri (L. reuteri), formerly Lactobacillus reuteri, is currently used in probiotic products.

The design of the study is based on the aim to study the safety and tolerability of a novel strain of the probiotic Limosilactobacillus reuteri (L. reuteri) in a limited number of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female subject aged 18-65 years inclusive.
3. Body Mass Index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2.
4. Clinically normal medical history, physical findings, vital signs, and laboratory values at the time of screening, as judged by the Investigator.
5. Female subjects of child bearing potential must practice abstinence (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose. Female subjects of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with simultaneous detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory).

Exclusion Criteria:

1. History of or ongoing clinically significant disease that, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the IP.
3. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the study.
5. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibodies or HIV.
6. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to Lactobacillus probiotic treatment.
7. History of, or ongoing GI disorder, including but not limited to irritable bowel syndrome (IBS), constipation, loose stools or excess gas which, in the discretion of the Investigator, may influence the results or the subject's ability to participate in the study.
8. Regular use of any prescribed or non-prescribed medication including antacids and analgesics within 2 weeks prior to the first administration of IP, at the discretion of the Investigator.
9. Any use of antibiotics (except local treatment, e.g., eye drops) within 2 weeks prior to the first administration of IP.
10. Regular use of supplements, i.e., tablets, drops, capsules etc, that contain L. reuteri or any other probiotics within 2 weeks prior to the first administration of IP.
11. Regular intake of foods or beverages that contain L. reuteri or any other probiotics, e.g., yoghurt and other probiotic dairy products, within 2 weeks prior to the first administration of IP. Foods that contain microorganisms, live or dead, that do not confer any health benefit on the host, e.g., regular yoghurt, are allowed.
12. Planned treatment or treatment with an investigational drug within 3 months prior to Day 1. Subjects consented and screened but not dosed in previous clinical studies are not excluded.
13. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times per week is allowed before the screening visit.
14. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IP. Drugs of abuse and alcohol will also be screened during the study (refer to Section 9.6.1).
15. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
16. Presence or history of drug abuse, as judged by the Investigator.
17. History of, or current use of, anabolic steroids, as judged by the Investigator.
18. Excessive caffeine consumption defined by a daily intake of > 5 cups of caffeine-containing beverages.
19. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the 3 months prior to screening.
20. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of treatment emergency adverse events (safety and tolerability). | 28 days
  The product to be investigated is a probiotic product and not an investigational medicinal product. However, the procedures for monitoring, collecting and reporting of AEs will be the same as for an investigational medicinal product.
  Vital signs, systolic and diastolic blood pressure and pulse will be measured. Vital signs will be judged as normal, abnormal, not clinically significant or abnormal, clinically significant.
  Safety laboratory parameters, blood samples for analysis of clinical chemistry and haematology will be analysed by routine analytical methods.
  Urine drug screen and urine pregnancy test will be performed. Abnormal values assessed by the Investigator as clinically significant will be reported as AEs. If an abnormal value is associated with corresponding clinical signs or symptoms, the sign/symptoms should be reported as the AE.

SECONDARY OUTCOMES:
To evaluate tolerability in terms of gastrointestinal symptoms | 28 days
  To evaluate gastrointestinal symptoms by using Gastrointestinal Symptom Rating Scale (GSRS) over the last week. The questionnaire will be answered by the subjects at visit 2 to 5.
  The Gastrointestinal Symptom Rating Scale is a disease-specific instrument. The 15 items are combined into five clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The subjects are asked to numerically score their subjective symptoms 1-7. Thus the lowest score is 15 and the highest is105. The higher score the worse outcome. The reliability and validity of the Gastrointestinal Symptom Rating Scale are well-documented, and norm values for a general population are available.
  The data collected using the Gastrointestinal Symptom Rating Scale does not constitute AEs and will not be reported as numerical results. Accordingly, no causality assessment by the Investigator will be performed for the Gastrointestinal Symptom Rating Scale questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein-Hedin, MD, Principal Investigator — CTC Clinical Trial Consultants AB,Dag Hammarskjolds v- 10B, SE-752 37 Uppsala, Sweden
Locations (2):
- Sweden (2):
  - Clinical Trial Consultants AB, Uppsala
  - CTC, Dag Hammarskjölds väg 10B, Uppsala